CLINICAL TRIAL: NCT02797327
Title: Molecular Signature of Karen and Burmese Pregnant Women on the Thailand-Myanmar Border
Brief Title: Molecular Signature Pregnancy
Acronym: MSP
Status: Completed | Type: Observational
Sponsor: University of Oxford (Other)
Collaborators: Sidra Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: SMRU1502
Record Dates: First submitted 2016-05-04; First posted 2016-06-13 (Estimated); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Pregnancy
Keywords: Molecular signature; Thailand-Myanmar border

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample, vaginal swab and stool specimen will be collected.
Oversight: Data Monitoring Committee: No

SUMMARY:
The primary goal of the study is to identify biomarkers from the molecular signature predictive of pre-term birth. This will be achieved through high frequency sampling and profiling throughout pregnancy.

DETAILED DESCRIPTION:
BACKGROUND Preterm birth occurs before 37 weeks and is a major cause of neonatal mortality and morbidity, and affecting 8% of newborns on the Thailand-Myanmar border. Identifying biochemical markers that are associated with preterm birth can guide in designing the most effective targeted intervention strategies for women at risk.

In order to identify biomarkers signatures predictive of preterm birth the investigators will employ high throughput profiling technologies (aka "a systems approach") that maximize the amount of information that can be obtained and knowledge generated from each participant sample. Preliminary data will also be obtained for infectious complications in order to assess potential for a systems approach such approach in detecting infectious events before onset of clinical symptoms or in absence of clinical symptoms. The rationale behind such approach and its importance for establishing personalized medicine approaches was detailed in a recent opinion article published. In addition parallel studies will be carried out in other countries such as Qatar and the US in order to assess environmental influences on blood and transcriptome signatures.

RESEARCH DESIGN This is a prospective pregnancy cohort from the first trimester until post-partum. The investigators are unable to predict which women will have preterm birth or infection.

STUDY POPULATION 400 Pregnant women with confirmed viable pregnancy of more than 8+0 weeks and less than 14 weeks of pregnancy, who are healthy, intend to deliver at SMRU and can attend for two weekly ANC visits.

METHOD AND TECHNIQUE

* Pregnant women attending SMRU ANC clinics will be invited to participate in the study.
* Study samples will include:

  1. A small blood volume (100 micro litres) will be collected by finger prick sampling via a capillary straw. The sample will be transferred into a microtube containing an RNA stabilizing solution and stored at -80°C. This will be repeated every two weeks, delivery and post-partum.
  2. A stool sample will be collected and stored at -80°C. This will be collected each trimester, delivery and post-partum.
  3. A vaginal swab will be collected from the posterior fornix under direct visualization by the midwife; and stored at -80°C. This will be collected each trimester, delivery and post-partum.

The post-partum visits, will be at 4-6 weeks and at 3months. The investigators estimate 15-18 blood samples, and 6 stool and vaginal swabs will be collected per women if they attend as expected. Fetal growth will be measured by 5-6 weekly ultrasound scans.

The sample set will be repeated if the woman has fever during pregnancy or post-partum (estimated at 5% of the women).

POTENTIAL VALUE Identifying biochemical markers that are associated with preterm can guide in designing the most effective targeted intervention strategies aimed at women at risk for preterm birth.

Funder & grant reference number: Sidra Medical and Research Center (Sidra)/ B9R01250; and supported by Wellcome [220211; assigned to Nicholas Day];

ELIGIBILITY:
Inclusion Criteria:

* Pregnant woman is willing and able to give informed consent for participation in the study.
* Karen or Burmese, age 18-49 years
* Healthy women with viable singleton first trimester (8+0 to < 14 weeks) pregnancy
* Plan to delivery at SMRU clinic
* Able (in the Investigators opinion) and willing to comply with all study requirements.

Exclusion Criteria:

The participant will not enter the study or continue in the study if ANY of the following apply:

* Emergency obstetric care required
* Pregnant woman (in the investigator's opinion) with medical or obstetrics complications which would make it difficult to comply with study requirements

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Target population: First trimester pregnant women with a viable pregnancy who will be followed for the outcome of interest of preterm births on the Thailand-Myanmar border
Sampling Method: Non-Probability Sample
Enrollment: 430 (Actual)
Dates: Start 2016-09-12 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
Characterization of the molecular signature of 30 preterm pregnancies defined by real-time PCR | up to 6 weeks post-partum

SECONDARY OUTCOMES:
Proportion of women who completed two weekly sampling | up to delivery
Proportion of rate of drop-out from sampling | up to delivery
Pain scores of the different samples from pregnant women. | up to 6 weeks post-partum
Molecular signature in relation to infection during pregnancy defined by real-time PCR | up to delivery
Molecular signature across the duration of pregnancy and post-partum time defined by real-time PCR | From enrolment at 8-14 weeks of pregnancy to 4-6 weeks post-partum

CONTACTS AND LOCATIONS:
Locations (1):
- Shoklo Malaria Research Unit, Mae Sot, Changwat Tak, Thailand

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Ahmad F, Lakshmanan AP, Alabduljabbar S, Ahmed SH, Ahmed A, Kabeer BSA, Marr AK, Kino T, Brummaier T, McGready R, Nosten F, Chaussabel D, Al Khodor S, Terranegra A. Placental and cord blood DNA methylation in preterm birth: exploring the epigenetic role of maternal dietary protein. NPJ Sci Food. 2025 Oct 14;9(1):206. doi: 10.1038/s41538-025-00566-w. PMID 41087373
- [Derived] Brummaier T, Syed Ahamed Kabeer B, Wilaisrisak P, Pimanpanarak M, Win AK, Pukrittayakamee S, Marr AK, Kino T, Al Khodor S, Terranegra A, Carrara VI, Nosten F, Utzinger J, Chaussabel D, Paris DH, McGready R. Cohort profile: molecular signature in pregnancy (MSP): longitudinal high-frequency sampling to characterise cross-omic trajectories in pregnancy in a resource-constrained setting. BMJ Open. 2020 Oct 10;10(10):e041631. doi: 10.1136/bmjopen-2020-041631. PMID 33040018
- [Derived] Brummaier T, Syed Ahamed Kabeer B, Lindow S, Konje JC, Pukrittayaamee S, Utzinger J, Toufiq M, Antoniou A, Marr AK, Suriyakan S, Kino T, Al Khodor S, Terranegra A, Nosten F, Paris DH, McGready R, Chaussabel D. A prospective cohort for the investigation of alteration in temporal transcriptional and microbiome trajectories preceding preterm birth: a study protocol. BMJ Open. 2019 Jan 15;9(1):e023417. doi: 10.1136/bmjopen-2018-023417. PMID 30782707